CLINICAL TRIAL: NCT05678348
Title: Early Phase I Window of Opportunity Biomarker and Safety Trial to Test Pyrimethamine as an Inhibitor of NRF2 in HPV-unrelated, Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Pyrimethamine as an Inhibitor of NRF2 in HPV-unrelated Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Tilde Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202302068
Record Dates: First submitted 2022-12-20; First posted 2023-01-10 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer; Cancer of the Head and Neck
Keywords: head and neck cancer; squamous cell carcinoma; NRF2; pyrimethamine; treatment resistance
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pyrimethamine (Experimental): Pyrimethamine will be taken by mouth at a dose of 50 mg once daily for 14 days (+/-2 days) with the last dose the day prior to surgery.
  Interventions: Drug: Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine — Patients will be instructed to take their dose at approximately the same time each day.
  Other Names: Daraprim

SUMMARY:
NRF2 activation, observed in up to 40% of head and neck squamous cell carcinoma (HNSCC) tumors, plays a critical role in tumor progression, metastasis, and radiation therapy resistance. The investigators have recently discovered that pyrimethamine (PYR) and its analogs have an inhibitory effect on NRF2 activity in vitro and in mouse models via inhibition of dihydrofolate reductase (DHFR).

Pyrimethamine is an established drug that has been used for decades for treatment of protozoan infections and malaria. A growing body of research shows that it has potential antitumor activity, however its activity on growing human tumors has not been previously studied. The primary efficacy goal of this study is to evaluate the activity of pyrimethamine on human tumors as demonstrated by inhibition of DHFR and downregulation of NRF2 pathway activity. On-target inhibition of DHFR by pyrimethamine results in the stabilization and increased protein expression of human DHFR.

The primary efficacy hypothesis of this study is that treatment with pyrimethamine will result in a 50% increase in DHFR protein within the tumor cells as measured by quantitative western blot analysis. Secondarily, among those tumors classified as NRF2-active on pre-treatment biopsy, the investigators hypothesize there will be a 50% reduction in NRF2 activity as measured by SureQuant targeted proteomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, locally advanced (Stage III-IV) head and neck squamous cell carcinoma (HNSCC) undergoing surgical-based treatment with curative intent that is HPV-unrelated disease, defined as SCC of the oral cavity, larynx, or hypopharynx, p16 negative SCC of the oropharynx.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3.0 K/cumm
  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 50 mL/min by Cockcroft-Gault
* Able to swallow study drug
* The effects of pyrimethamine on the developing human fetus are unknown. For this reason and because it is in Pregnancy Category C, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.
* Patient must be able to undergo a research biopsy prior to starting treatment, or have previously banked baseline tumor biopsy of at least 20 mg of frozen tissue collected under Tissue Acquisition Protocol (IRB 201102323).

Exclusion Criteria:

* Prior therapy for this cancer.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Prior treatment with pyrimethamine in the year prior to HNSCC diagnosis.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pyrimethamine or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, current use of systemic immunosuppressive medications, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Documented megaloblastic anemia due to folate deficiency.
* Treatment with anticoagulant or antiplatelet therapy in the year prior to HNSCC diagnosis.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of Day 1.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Active alcohol abuse in the opinion of the treating physician.
* Currently taking phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Change in Log2 of tumor DHFR expression as measured by western blot analysis | Pre-treatment and post-treatment (estimated to be 14 days)

SECONDARY OUTCOMES:
Safety and tolerability of pyrimethamine as measured by number of adverse events | From start of treatment through Day 43 (estimated to be 6 weeks)
Change in Log2 of NRF2 activity score as measured using the NRF2 SureQuant proteomic assay | Pre-treatment and post-treatment (estimated to be 14 days)
Number of grade 3 or higher adverse events due to pyrimethamine | From start of treatment through Day 43 (estimated to be 6 weeks)
Number of participants with a delay in surgery by ≥ 10 days due to pyrimethamine | Through completion of follow-up (estimated to be 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Zolkind, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu